CLINICAL TRIAL: NCT02987985
Title: Efficacy of Opioid-free Anesthesia in Reducing Postoperative Respiratory Depression in Children Undergoing Tonsillectomy: a Pilot Study
Brief Title: Efficacy of Opioid-free Anesthesia in Reducing Postoperative Respiratory Depression in Children Undergoing Tonsillectomy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Saskatchewan (Other)
Responsible Party: Principal Investigator, Jonathan Gamble, Principle Investigator, University of Saskatchewan
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: BIO 16-255
Record Dates: First submitted 2016-11-29; First posted 2016-12-09 (Estimated); Last update posted 2021-08-10 (Actual); Status verified 2021-08

CONDITIONS: Anesthesia; General Anesthesia; Analgesics, Opioid; Postoperative Complications; Pathologic Processes; Physiologic Effects of Drugs; Narcotics; Analgesics; Sleep Disordered Breathing; Obstructive Sleep Apnea of Child; Tonsillectomy; Respiratory Depression; Dexmedetomidine; Ketamine; Lidocaine; Gabapentin; Pulse Oximetry
Keywords: Opioid-sparing; Opioid-free
MeSH Terms: conditions — Postoperative Complications; Pathologic Processes; Sleep Apnea Syndromes; Respiratory Insufficiency | interventions — Acetaminophen; Gabapentin; Ketamine; Lidocaine; Dexmedetomidine; Fentanyl; Dexamethasone; Ondansetron; Sevoflurane

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Opioid-free anesthesia (Experimental): Opioid-free preoperative medications, Opioid-free pre-intubation medications, Opioid-free maintenance medication, postoperative nausea and vomiting prophylaxis
  Interventions: Drug: Acetaminophen, gabapentin; Drug: Ketamine , Lidocaine , Dexmedetomidine; Drug: Dexamethasone , Ondansetron; Drug: Sevoflurane
- Opioid-sparing anesthesia (Active Comparator): Opioid-sparing preoperative medications, Opioid sparing pre-intubation medications, Opioid-sparing maintenance medications, postoperative nausea and vomiting prophylaxis
  Interventions: Drug: Acetaminophen; Drug: Fentanyl, Dexmedetomidine; Drug: Dexamethasone , Ondansetron; Drug: Sevoflurane, Fentanyl

INTERVENTIONS:
Drug: Acetaminophen, gabapentin — acetaminophen 15 mg/kg, gabapentin 10 mg/kg
  Other Names: Opioid-free preoperative medications
  Arms: Opioid-free anesthesia
Drug: Acetaminophen — acetaminophen 15 mg/kg
  Other Names: Opioid-sparing preoperative medications
  Arms: Opioid-sparing anesthesia
Drug: Ketamine , Lidocaine , Dexmedetomidine — Ketamine 0.5 mg/kg, Lidocaine 1 mg/kg, Dexmedetomidine 0.3 mcg/kg
  Other Names: Opioid-free pre-intubation medications
  Arms: Opioid-free anesthesia
Drug: Fentanyl, Dexmedetomidine — Fentanyl 0.5 mcg/kg, Dexmedetomidine 0.3 mcg/kg
  Other Names: Opioid sparing pre-intubation medications
  Arms: Opioid-sparing anesthesia
Drug: Dexamethasone , Ondansetron — Dexamethasone 150 mcg/kg, Ondansetron 50 mg/kg
  Other Names: Postoperative nausea and vomiting prophylaxis
Drug: Sevoflurane — Sevoflurane (dose titrated to effect)
  Other Names: Opioid-free maintenance medication
  Arms: Opioid-free anesthesia
Drug: Sevoflurane, Fentanyl — Sevoflurane (dose titrated to effect), Fentanyl as needed (dose at anesthesiologist's discretion)
  Other Names: Opioid-sparing maintenance medications
  Arms: Opioid-sparing anesthesia

SUMMARY:
The objective of this trial is to determine whether an opioid-free general anesthetic (OFA) technique utilizing ketamine, dexmedetomidine, lidocaine, and gabapentin can help reduce postoperative respiratory depression in the post-anesthesia care unit and ward in children with sleep-disordered breathing undergoing tonsillectomy when compared with traditional opioid-containing techniques. It is expected that this OFA regimen will have a measurable reduction on postoperative respiratory depression in children with sleep-disordered breathing.

DETAILED DESCRIPTION:
The objective of this trial is to determine whether an opioid-free general anesthetic can help reduce postoperative respiratory depression in the post-anesthesia care unit and ward in children with sleep-disordered breathing undergoing tonsillectomy when compared with traditional opioid-containing techniques.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 0-12 years with Sleep Disordered Breathing (SDB) who are scheduled for elective Tonsillectomy/AdenoTonsillectomy (T/AT) will be recruited at Royal University Hospital, Saskatoon, Saskatchewan.

Exclusion Criteria:

* age > 12; American Society of Anesthesiologists (ASA) Classification > IV; significant cardiorespiratory, neurological, craniofacial, hepatic, renal, or genetic disorders, excluding SDB; concomitant surgical procedures other than myringotomy and tubes; and allergy to any of the study drugs

Max Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 2017-10-15 (Actual); Primary Completion 2019-09-20 (Actual); Study Completion 2020-12-20 (Actual)

PRIMARY OUTCOMES:
Respiratory depression | 24 hours following surgery
  Number of desaturation events (oxygen saturation by pulse oximetry (SPO2) <90%) as measured by a Masimo Radical-7 pulse oximeter during the first postoperative night's sleep

SECONDARY OUTCOMES:
Quantified opioid consumption | 24 hours following surgery
  Quantified opioid consumption
Pediatric Agitation Emergence Delirium (PAED) scale | 24 hours following surgery
  Pediatric Agitation Emergence Delirium (PAED) scale
Face Legs Activity Cry Consolability (FLACC) scale | 24 hours following surgery
  Face Legs Activity Cry Consolability (FLACC) scale
Time until Post Anesthesia Care Unit (PACU) discharge readiness | 24 hours following surgery
  Time until Post Anesthesia Care Unit (PACU) discharge readiness
Other adverse effects | 24 hours following surgery
  Other adverse effects

CONTACTS AND LOCATIONS:
Overall Officials: Jon Gamble, MD, Principal Investigator — University of Saskatchewan
Locations (1):
- Royal University Hospital, Saskatoon, Saskatchewan, Canada

IPD SHARING:
Plan to Share IPD: No